CLINICAL TRIAL: NCT04470583
Title: Evaluation of Clinical Parameters Following COVID-19 Infection in Pregnancy (COpregVID)
Brief Title: Evaluating Clinical Parameters of COVID-19 in Pregnancy
Acronym: COpregVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W20/034; 283995 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; 2019 Novel Coronavirus Infection; COVID-19 Infection
Keywords: COVID-19; Pregnancy; Retrospective case review
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild/moderate COVID-19 affected pregnant and postnatal women: Pregnant and postnatal women who contracted COVID-19 and recovered without the need for ventilation will be classified as mild to moderate. Participants will be aged between 18-50 years old.
- Severe/Critical COVID-19 affected pregnant and postnatal women: Pregnant and postnatal women who are admitted to hospital after contracting COVID-19 and received ventilatory support before recovering will be classified as severe to critical. Participants will be aged between 18-50 years old.
  These participants will be identified from Intensive Treatment Unit (ITU), and standard COVID-19 wards.
- Mild/moderate COVID-19 affected non-pregnant participants: Both male and non-pregnant female participants who contracted COVID-19 and recovered without the need for ventilation will be classified as mild to moderate. Participants will be aged between 18-60 years old.
- Severe/Critical COVID-19 affected non-pregnant participants: Both male and non-pregnant female participants who are admitted to hospital after contracting COVID-19 and received ventilatory support before recovering will be classified as severe to critical. Participants will be aged between 18-60 years old. These participants will be identified from Intensive Treatment Unit (ITU), and standard COVID-19 wards.

SUMMARY:
Coronavirus infection, also known as COVID-19, has become a global pandemic with over 3 million cases and 250,000 deaths worldwide. Coronaviruses (CoV) belong to a family of viruses that predominately infect mammals and birds, affecting their lungs, intestinal tract, liver and nervous systems. Prior to the discovery of the current novel coronavirus strain (SARS-CoV-2), there were six different strains that are known to infect humans, which includes the virus that caused the severe acute respiratory syndrome (SARS) pandemic in 2002. In humans, the majority of severe illness from SARs and COVID-19 is due to inflammation of the lungs and pneumonia. Pregnancy poses a significantly increased risk of viral pneumonia and during SARS more pregnant women required intensive care and breathing support, and the proportion of deaths was higher when compared to non-pregnant adults. Furthermore, kidney failure and development of abnormal blood clotting disorders, which occurs during severe infection, is more common in pregnancy and the associated changes in blood vessels extend to the placentas of infected pregnant women, thus potentially affecting the fetus. This makes pregnant women affected by the virus at high risk of developing severe complications. Fortunately, there have been a number of biomarkers identified that are associated with illness severity. These include, specialised white blood cells, blood clotting cells and constituents, as well as other measures of heart and kidney function. We propose that these biomarkers are important correlates of clinical disease severity and prognosis in pregnant and postnatal women. This knowledge has the potential to help clinicians during this pandemic to better manage and care for their patients.

DETAILED DESCRIPTION:
This study will be a retrospective case review using existing clinical data from participating centres. To date there have already been 18,000 confirmed cases in Greater London. Our study design will aim to include patients who were diagnosed with COVID-19 at the start of the pandemic as well as new and current cases.

The study design requires data to be extracted from National Health Service (NHS) electronic and paper notes, which will contain patient identifiable information. For confidentiality, all patient identifiable data will only be collected by members of the direct care team. This data will be encrypted and stored in a local NHS trust computer at participating sites. In order to maintain confidentiality, all data will then be anonymised before being inputted on a data collection tool and spreadsheet. Therefore, research teams will only be provided with a de-identified dataset. This data will be transferred across to the study co-ordination centre, following NHS information governance rules for data to be compiled and analysed. At the co-ordination centre, this data will be stored in an Imperial College London computer, and will only be accessible to the research team.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection
* 18-50 years for Groups A and B and 18-60 years for Groups C and D
* Female for groups A and B. Both male and female for groups C and D.

Exclusion Criteria:

* Participants who have previously been part of a SARS-CoV-2 vaccine trial.
* Current hospital admission due to another respiratory disease, such as influenza.
* Obvious clinical deterioration due to another medical problem such as cardiovascular disease, diabetes or malignancy.
* Evidence of HIV infection and/or participants on anti-retroviral drug therapy.
* Participants on chemotherapy, biologics, immune-modulators or immunosuppressive drugs (not including intramuscular steroids for fetal lung maturity).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Due to the novel nature of this project, patients will not be stratified for specific demographic differences such as age, ethnicity or BMI. As there is very little data on SARS or COVID-19 infection in pregnant and postnatal women within 6 weeks of birth, power calculations used data from non-pregnant cases. In our institution so far, we have had 17 pregnant or postnatal women with COVID-19, and approximately 5 non-pregnant women of childbearing age out of a total of 273 cases (as of 1nd May 2020). Therefore, for some of non-pregnant data collection, we will be using data obtained from both male and female participants with a wider age range than our pregnant and postnatal group. Once all the data has been collected, we may stratify them based on age, gender, BMI, and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12-02 (Estimated)

PRIMARY OUTCOMES:
Proportions of leukocyte subsets and thrombocytes in pregnant/postnatal and non-pregnant COVID-19 positive women. | From the start of the study up until one month prior to study end.
  Data collection and analysis on the proportions of leukocyte subsets and thrombocytes in pregnant/postnatal and non-pregnant COVID-19 positive patients during acute infection and recovery.
Concentrations of other biochemical markers of severity in pregnant and non-pregnant COVID-19 positive women. | From the start of the study up until one month prior to study end.
  Data collection and analysis on the concentrations of other biochemical markers of severity in pregnant and non-pregnant COVID-19 positive patients during acute infection and recovery.

SECONDARY OUTCOMES:
Profiling of clinical severity, determined by clinical symptoms and observations in pregnant and non-pregnant COVID-19 positive women. | From the start of the study up until one month prior to study end.
  Data collection and analysis on profiling of clinical severity, determined by clinical symptoms and observations in pregnant and non-pregnant COVID-19 positive women.

CONTACTS AND LOCATIONS:
Overall Officials: Nishel Shah, MRCOG, PhD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No
Research team wishes to enable any meta-analyses of COVID-19 trials making appropriate requests. No plan to share IPD has been made at this time.

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Wevers BA, van der Hoek L. Recently discovered human coronaviruses. Clin Lab Med. 2009 Dec;29(4):715-24. doi: 10.1016/j.cll.2009.07.007. PMID 19892230
- [Background] Masters PS. The molecular biology of coronaviruses. Adv Virus Res. 2006;66:193-292. doi: 10.1016/S0065-3527(06)66005-3. PMID 16877062
- [Background] van der Hoek L, Pyrc K, Jebbink MF, Vermeulen-Oost W, Berkhout RJ, Wolthers KC, Wertheim-van Dillen PM, Kaandorp J, Spaargaren J, Berkhout B. Identification of a new human coronavirus. Nat Med. 2004 Apr;10(4):368-73. doi: 10.1038/nm1024. Epub 2004 Mar 21. PMID 15034574
- [Background] Sahu KK, Mishra AK, Lal A. Coronavirus disease-2019: An update on third coronavirus outbreak of 21st century. QJM. 2020 May 1;113(5):384-386. doi: 10.1093/qjmed/hcaa081. No abstract available. PMID 32125418
- [Background] Petrosillo N, Viceconte G, Ergonul O, Ippolito G, Petersen E. COVID-19, SARS and MERS: are they closely related? Clin Microbiol Infect. 2020 Jun;26(6):729-734. doi: 10.1016/j.cmi.2020.03.026. Epub 2020 Mar 28. PMID 32234451
- [Background] Yang M, Ng MH, Li CK. Thrombocytopenia in patients with severe acute respiratory syndrome (review). Hematology. 2005 Apr;10(2):101-5. doi: 10.1080/10245330400026170. PMID 16019455
- [Background] He WQ, Chen SB, Liu XQ, Li YM, Xiao ZL, Zhong NS. [Death risk factors of severe acute respiratory syndrome with acute respiratory distress syndrome]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2003 Jun;15(6):336-7. Chinese. PMID 12837163
- [Background] Wong RS, Wu A, To KF, Lee N, Lam CW, Wong CK, Chan PK, Ng MH, Yu LM, Hui DS, Tam JS, Cheng G, Sung JJ. Haematological manifestations in patients with severe acute respiratory syndrome: retrospective analysis. BMJ. 2003 Jun 21;326(7403):1358-62. doi: 10.1136/bmj.326.7403.1358. PMID 12816821
- [Background] Lippi G, Plebani M, Henry BM. Thrombocytopenia is associated with severe coronavirus disease 2019 (COVID-19) infections: A meta-analysis. Clin Chim Acta. 2020 Jul;506:145-148. doi: 10.1016/j.cca.2020.03.022. Epub 2020 Mar 13. PMID 32178975
- [Background] Xu P, Zhou Q, Xu J. Mechanism of thrombocytopenia in COVID-19 patients. Ann Hematol. 2020 Jun;99(6):1205-1208. doi: 10.1007/s00277-020-04019-0. Epub 2020 Apr 15. PMID 32296910
- [Background] Fogarty H, Townsend L, Ni Cheallaigh C, Bergin C, Martin-Loeches I, Browne P, Bacon CL, Gaule R, Gillett A, Byrne M, Ryan K, O'Connell N, O'Sullivan JM, Conlon N, O'Donnell JS. COVID19 coagulopathy in Caucasian patients. Br J Haematol. 2020 Jun;189(6):1044-1049. doi: 10.1111/bjh.16749. Epub 2020 May 17. PMID 32330308
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Mar 27;5(1):33. doi: 10.1038/s41392-020-0148-4. No abstract available. PMID 32296069
- [Background] Fan BE, Chong VCL, Chan SSW, Lim GH, Lim KGE, Tan GB, Mucheli SS, Kuperan P, Ong KH. Hematologic parameters in patients with COVID-19 infection. Am J Hematol. 2020 Jun;95(6):E131-E134. doi: 10.1002/ajh.25774. Epub 2020 Mar 19. No abstract available. PMID 32129508
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zheng HY, Zhang M, Yang CX, Zhang N, Wang XC, Yang XP, Dong XQ, Zheng YT. Elevated exhaustion levels and reduced functional diversity of T cells in peripheral blood may predict severe progression in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):541-543. doi: 10.1038/s41423-020-0401-3. Epub 2020 Mar 17. No abstract available. PMID 32203186
- [Background] Giamarellos-Bourboulis EJ, Netea MG, Rovina N, Akinosoglou K, Antoniadou A, Antonakos N, Damoraki G, Gkavogianni T, Adami ME, Katsaounou P, Ntaganou M, Kyriakopoulou M, Dimopoulos G, Koutsodimitropoulos I, Velissaris D, Koufargyris P, Karageorgos A, Katrini K, Lekakis V, Lupse M, Kotsaki A, Renieris G, Theodoulou D, Panou V, Koukaki E, Koulouris N, Gogos C, Koutsoukou A. Complex Immune Dysregulation in COVID-19 Patients with Severe Respiratory Failure. Cell Host Microbe. 2020 Jun 10;27(6):992-1000.e3. doi: 10.1016/j.chom.2020.04.009. Epub 2020 Apr 21. PMID 32320677
- [Background] Kong WH, Li Y, Peng MW, Kong DG, Yang XB, Wang L, Liu MQ. SARS-CoV-2 detection in patients with influenza-like illness. Nat Microbiol. 2020 May;5(5):675-678. doi: 10.1038/s41564-020-0713-1. Epub 2020 Apr 7. PMID 32265517
- [Background] Wong SF, Chow KM, Leung TN, Ng WF, Ng TK, Shek CC, Ng PC, Lam PW, Ho LC, To WW, Lai ST, Yan WW, Tan PY. Pregnancy and perinatal outcomes of women with severe acute respiratory syndrome. Am J Obstet Gynecol. 2004 Jul;191(1):292-7. doi: 10.1016/j.ajog.2003.11.019. PMID 15295381
- [Background] LoMauro A, Aliverti A. Respiratory physiology of pregnancy: Physiology masterclass. Breathe (Sheff). 2015 Dec;11(4):297-301. doi: 10.1183/20734735.008615. PMID 27066123
- [Background] Zollner J, Howe LG, Edey LF, O'Dea KP, Takata M, Gordon F, Leiper J, Johnson MR. The response of the innate immune and cardiovascular systems to LPS in pregnant and nonpregnant mice. Biol Reprod. 2017 Aug 1;97(2):258-272. doi: 10.1093/biolre/iox076. PMID 29044422
- [Background] Schwartz DA, Graham AL. Potential Maternal and Infant Outcomes from (Wuhan) Coronavirus 2019-nCoV Infecting Pregnant Women: Lessons from SARS, MERS, and Other Human Coronavirus Infections. Viruses. 2020 Feb 10;12(2):194. doi: 10.3390/v12020194. PMID 32050635
- [Background] Cerbulo-Vazquez A, Figueroa-Damian R, Arriaga-Pizano LA, Hernandez-Andrade E, Mancilla-Herrera I, Flores-Mejia LA, Arteaga-Troncoso G, Lopez-Macias C, Isibasi A, Mancilla-Ramirez J. Pregnant women infected with pandemic H1N1pdm2009 influenza virus displayed overproduction of peripheral blood CD69+ lymphocytes and increased levels of serum cytokines. PLoS One. 2014 Sep 25;9(9):e107900. doi: 10.1371/journal.pone.0107900. eCollection 2014. PMID 25254368
- [Background] Du RH, Liang LR, Yang CQ, Wang W, Cao TZ, Li M, Guo GY, Du J, Zheng CL, Zhu Q, Hu M, Li XY, Peng P, Shi HZ. Predictors of mortality for patients with COVID-19 pneumonia caused by SARS-CoV-2: a prospective cohort study. Eur Respir J. 2020 May 7;55(5):2000524. doi: 10.1183/13993003.00524-2020. Print 2020 May. PMID 32269088
- [Background] Han Y, Zhang H, Mu S, Wei W, Jin C, Tong C, Song Z, Zha Y, Xue Y, Gu G. Lactate dehydrogenase, an independent risk factor of severe COVID-19 patients: a retrospective and observational study. Aging (Albany NY). 2020 Jun 24;12(12):11245-11258. doi: 10.18632/aging.103372. Epub 2020 Jun 24. PMID 32633729
- [Background] ICNARC report on COVID-19 in critical care London, UK: Intensive Care National Audit & Research Centre (ICNARC); 2020 04 April 2020.
- [Background] Bouch, D. C., & Thompson, J. P. (2008). Severity scoring systems in the critically ill. Continuing Education in Anaesthesia Critical Care & Pain, 8(5), 181-185. https://doi.org/10.1093/bjaceaccp/mkn033
- [Background] Zhang G, Hu C, Luo L, Fang F, Chen Y, Li J, Peng Z, Pan H. Clinical features and short-term outcomes of 221 patients with COVID-19 in Wuhan, China. J Clin Virol. 2020 Jun;127:104364. doi: 10.1016/j.jcv.2020.104364. Epub 2020 Apr 9. PMID 32311650
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Greer O, Shah NM, Johnson MR. Maternal sepsis update: current management and controversies. The Obstetrician & Gynaecologist. 2020;22(1):45-55.
- [Background] Zheng Y, Huang Z, Ying G, Zhang X, Ye W, Hu Z, et al. Study of the lymphocyte change between COVID-19 and non-COVID-19 pneumonia cases suggesting other factors besides uncontrolled inflammation contributed to multi-organ injury. medRxiv. 2020:2020.02.19.20024885.
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- See also: The World Health Organisation's advice and guidance on the coronavirus disease (COVID-19) pandemic — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: The UK Government's report on the number of coronavirus (COVID-19) cases and risk in the UK — http://www.gov.uk/guidance/coronavirus-covid-19-information-for-the-public
- See also: The economic consequences of Covid-19 ' an article by Iain Begg, Professor at the London School of Economics and Political Science — http://blogs.lse.ac.uk/europpblog/2020/04/06/the-economic-consequences-of-covid-19/